CLINICAL TRIAL: NCT04606329
Title: A Multicenter, Randomized, Open-label, Parallel Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of LuminoMark Inj. Versus Charcotrace Inj. in Patients With Nonpalpable Breast Lesions
Brief Title: To Evaluate the Efficacy and Safety of LuminoMark Injection in Patients With Nonpalpable Breast Lesions(Phase 3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HL_LMN_301
Record Dates: First submitted 2020-10-14; First posted 2020-10-28 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Breast Diseases
Keywords: Nonpalpable Breast Lesions
MeSH Terms: conditions — Breast Diseases | interventions — Fluorescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LuminoMark inj. (Experimental): Injection LuminoMark inj. 0.2mL once in this study.
  Interventions: Drug: LuminoMark inj.(Conc. for fluorescence)
- Charcotrace Inj. (Active Comparator): Charcotrace Inj. about 0.3~1mL
  Interventions: Drug: Charcotrace Inj.

INTERVENTIONS:
Drug: LuminoMark inj.(Conc. for fluorescence) — Injection LuminoMark inj. (Conc. for fluorescence) 0.2mL once in this study.
  Arms: LuminoMark inj.
Drug: Charcotrace Inj. — Injection Charcotrace Inj. about 0.3~1mL once in this study.
  Arms: Charcotrace Inj.

SUMMARY:
This study is a multicenter, Randomized, Open-label, Parallel, Phase 3 Clinical Trial in 8 weeks for screening, once Investigational product injection, Follow up visit.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of LuminoMark inj. (Conc. for fluorescence) localization in patients with nonpalpable breast lesions.

ELIGIBILITY:
Inclusion Criteria:

1. 19 years ≤ age ≥ 80 years
2. Those who have lesion vial mammography and breast ultrasound
3. Those who be expected to do operation about non palpable breast lesion excision
4. Written consent voluntarily to participate in this clinical trial

Exclusion Criteria:

1. Patients who be expected to do mastectomy
2. Patients with multiple tumor or diffuse microcalcification
3. Patients who have ink on invasive cancer or ductal carcinoma in situ despite 3 times local resection
4. Patients who were treated with moderate to severe radiotherapy
5. Patients who were treated with neoadjuvant Chemotherapy
6. Patients with active invading skin connective tissue disease
7. Patients with local progressing breast cancer or inflammatory local progressing breast cancer
8. Patients who have an allergy to investigational product or any of the component with the Investigational product
9. Patients who disagree about contraception for this clinical trial
10. A pregnant women or lactating women
11. Patients who participated in other clinical trials within the past 12 weeks from the date of informed consent
12. Patients who investigators determines unsuitable for this clinical trial

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-01-28 (Actual)

PRIMARY OUTCOMES:
Negative Resection margin rate | Visit 5 (Day 14 ~Day 24)
  The presence or absence of margin involvement in the resected breast lesions

SECONDARY OUTCOMES:
Technical success rate | Visit 3 (Day 0)
  The proportion of colored lesion when make an incision
Coloring confirmation rate of excision lesion | Visit 3 (Day 0)
  The proportion of colored excision lesion
Pathologic perfection | Visit 5 (Day 14 ~Day 24)
  Pathologic perfection is how well the surgeon removed the lesion compared to an identified by gross pathologic method. Visit 5, Investigators calculate 'Pathologic perfection' using by the formula. This formula's calculation method is as follows. [Pathologic perfection = the longest diameter of measured lesion by gross(=visual) pathologic method / the longest diameter of removed lesion after surgery]
Pigmentation rate | Visit 5 (Day 14 ~Day 24)
  Check whether skin is pigmented or not
Re-operation rate | Visit 5 (Day 14 ~Day 24)
  The number of subjects who need re-operation is evaluated based on the investigator's comprehensive judgment including histopathology test results.
Procedure complication rate | Visit 4, 5 (Day 1, Day 14 ~Day 24)
  Evaluate the numbers of subjects with procedure complication after lesion removal

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea